CLINICAL TRIAL: NCT02177149
Title: Mobile Computing Platform to Improve Outcomes From Deep Brain Stimulation Therapy
Brief Title: Nurse Management of Neuromodulation Therapy
Acronym: DBS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is no longer at MCW, study has been closed
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Christopher Butson, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB_00078062
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Parkinson's
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): DBS using standard of care.
  Interventions: Device: Standard of Care
- DBS Clinical Support System (Experimental): DBS using Clinical Support System.
  Interventions: Device: DBS using Clinical Support System.

INTERVENTIONS:
Device: Standard of Care — Patients in the standard of care arm will have their DBS programmed per standard of care which is testing multiple settings and looking for symptom relief through a trial and error process.
  Arms: Standard of Care
Device: DBS using Clinical Support System. — The DBS RN (Registered Nurse) will use ImageVis3D Mobile app on the iPad to program the DBS system, this software does not interact with imaging systems. The study team uses identified images provided by the Froedtert PACS system, de identifies them, adds a study code. The images are loaded into the software system and used to identify the leads locations. The Patients will be assessed for 6 months starting with the initial DBS programming session. Importantly, the investigators do not anticipate that the clinical decision support tool will provide the final DBS settings, nor do the investigators anticipate that the approach will obviate the need for motor exams. The clinical decision support system will help nurses choose good initial settings and then explore around those initial settings.
  Arms: DBS Clinical Support System

SUMMARY:
The central hypothesis is that the use of a DBS (Deep Brain Stimulation) clinical decision support system for individual patient management will enable considerable time savings compared to standard care. This hypothesis was formulated from pilot studies that showed dramatic decreases in DBS programming time compared to standard care for clinicians who used an iPad-based decision support system (99% time savings from over 4 hours to 2 minutes. Study group Parkinson's patients with DBS Systems

DETAILED DESCRIPTION:
In most cases these subjects have failed to maintain adequate control of their symptoms on medications alone.

The Diagnosis of PD (Parkinson's Disease) and the decision to have DBS qualifies a subject for enrollment. Subjects would be selected because they will require DBS programming.

The investigators will prospectively enroll 20 PD DBS patients at the Froedtert Movement Disorders Center (surgical targets: subthalamic nucleus (STN) or internal segment of globus pallidus (GPi). Post-operative care, patients will be randomized 1/1 to standard care or using the clinical decision support system. The DBS RN will use ImageVis3D Mobile app on the iPad to program the DBS system, this software does not interact with Froedtert imaging systems. The study team uses identified images provided by the Froedtert PACS system, de identifies them, adds a study code. The images are loaded into the software system and used to identify the leads locations. The Patients will be assessed for 6 months starting with the initial DBS programming session. Importantly, the investigators do not anticipate that the clinical decision support tool will provide the final DBS settings, nor do we anticipate that this approach will obviate the need for motor exams. The clinical decision support system will help nurses choose good initial settings and then explore around those initial settings.

The investigators will measure the time spent on DBS programming for patients in each group. The investigators will capture programming session duration, number of programming sessions and total time spent on DBS programming. The investigators will compare total time spent programming for the standard care versus the intervention group.

ELIGIBILITY:
Inclusion Criteria:

Subjects 18 and older with a diagnosis of Parkinson's Disease that are scheduled for Deep Brain Stimulation for control of their symptoms and are seen at the Froedtert Neurology Outpatient Clinic.

Exclusion Criteria:

Patient's that are not candidates for Deep Brain Stimulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Measure the effectiveness of DBS decision support system in an established clinic. | 6 months
  Patients will be assessed using the Unified Parkinson's Disease Rating Scale (UPDRS, motor section) by a blinded rater (Dr. Hiner, movement disorders neurologist). Patients will be tested in their best "On" state (e.g.on medication, on stimulation). The investigators will compare UPDRS-III scores for the standard care versus the intervention group. The UPDRS, Motor section is performed at each visit.
  Patient-Reported Outcomes
  The study team will capture patient-reported QOL (Quality of Life) using PDQ-39 (Parkinson 's Disease Questionnaire. The PDQ-39 is a validated, widely used scale completed by the patient, and is used to assess health-related quality of life in this cohort (Jenkinson, Peto, Fitzpatrick, Greenhall, & Hyman, 1995). Patients will fill out rating scales using a web-based form on an iPad or workstation during each clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Butson, PhD, Principal Investigator — Medical College of Wiscosnisn